CLINICAL TRIAL: NCT00759538
Title: Effect of Early Pulmonary Rehabilitation After Lung Transplantation in Patients With a Prolonged Length of Stay on the Waiting List and Hospitalization After Transplantation
Brief Title: Effect of Early Pulmonary Rehabilitation After Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Klinik Fallingbostel Rehabilitation Center (Unknown)
Responsible Party: Principal Investigator, Martin G Dierich, MD, MD, Hannover Medical School
Other Study IDs: MHH-2008-4
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Lung Transplantation
Keywords: Lung Transplantation; Pulmonary Rehabilitation; Exercise tolerance; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: lung transplant patients performing a three week lasting rehabilitation program

SUMMARY:
The purpose of this observation study is to evaluate the effects of an early, 3 week lasting rehabilitation program, that starts roundabout 4 weeks after lung or combined lung transplantation, on physical activity, functional and physical condition (6-min-walk, FEV1, ADL-score) and quality of life (SF36) in lung transplant recipients with a different length of stay on the waiting list and a different duration of hospitalization in the transplantation centre after transplantation.

DETAILED DESCRIPTION:
To which extend a prolonged duration from listing for lung transplantation until a successful transplantation or a long length of hospitalization may influence the success of a pulmonary rehabilitation, that starts after discharge from the transplantation centre, is still unknown.

Long waiting periods before transplantation and surgical, infectious or immunological complications after transplantation influence the physical condition and the quality of life of the organ recipient.

A poor physical condition before transplantation results in an unfavourable outcome in the first 12 months after transplantation.

At present it is unclear, whether a structured pulmonary rehabilitation may overwhelm differences between patients with a prolonged course roundabout the transplantation compared or not. At present it is not clear whether it is necessary for lung transplant recipients to participate in a rehabilitation program including structured exercise training.

The aim of this observational study is to assess the effect of a short-term pulmonary rehabilitation, that starts immediately after discharge from the transplantation centre on patients with a prolonged waiting period or an extended postoperative hospitalization.

* Hypothesis: a structured pulmonary rehabilitation early after transplantation may overwhelm poor physical and functional conditions after a prolonged period on the transplant waiting listor a prolonged hospitalization after transplantation resulting in a significant improvement in all transplanted patients
* Antithesis: a prolonged period on the waiting list before transplantation or a prolonged hospitalization after transplantation can not be influenced significantly by an early transplant rehabilitation resulting in a persistent lack of functional status and quality of life compared with a short waiting period or a normal duration of hospitalization after transplantation.
* Outcomes: functional status (6-min. walk, exercise capacity, FEV1, ADL), and quality of life (SF36) will be assessed at the beginning and on discharge from the rehabilitation centre.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of single or double lung transplants
* Recipients of combined (heart and lung or heart an liver) transplants

Ages: 17 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: lung transplant patients performing a three week lasting rehabilitation program
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-07; Primary Completion 2007-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Exercise capacity at the end of an early short-term after lung transplantation | 3 years

SECONDARY OUTCOMES:
Lung function | 3 years
Body composition | 3 years
Activities of daily living | 3 years
Health Status (SF-36) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dierich, MD, Principal Investigator — Hannover Medical School, Dpt. of Respiratory Medicine
Locations (1):
- Hannover Medical School, Dpt. of Respiratory Medicine, Hanover, Germany

REFERENCES:
- [Background] Tegtbur U, Sievers C, Busse MW, Pethig K, Warnecke G, Kugler C, Gutzlaff E, Kunsebeck HW, Struber M, Haverich A, Niedermeyer J. [Quality of life and exercise capacity in lung transplant recipients]. Pneumologie. 2004 Feb;58(2):72-8. doi: 10.1055/s-2003-812526. German. PMID 14961434
- [Background] Schwaiblmair M, Reichenspurner H, Muller C, Briegel J, Furst H, Groh J, Reichart B, Vogelmeier C. Cardiopulmonary exercise testing before and after lung and heart-lung transplantation. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1277-83. doi: 10.1164/ajrccm.159.4.9805113. PMID 10194177
- [Background] Schultz K, Bergmann KC, Kenn K, Petro W, Heitmann RH, Fischer R, Lang SM. [Effectiveness of inpatient pulmonary rehabilitation (AHB). Results of a multicenter prospective observation study]. Dtsch Med Wochenschr. 2006 Aug 18;131(33):1793-8. doi: 10.1055/s-2006-949155. German. PMID 16902901
- [Background] Maury G, Langer D, Verleden G, Dupont L, Gosselink R, Decramer M, Troosters T. Skeletal muscle force and functional exercise tolerance before and after lung transplantation: a cohort study. Am J Transplant. 2008 Jun;8(6):1275-81. doi: 10.1111/j.1600-6143.2008.02209.x. Epub 2008 Apr 29. PMID 18444941
- [Derived] Dierich M, Tecklenburg A, Fuehner T, Tegtbur U, Welte T, Haverich A, Warnecke G, Gottlieb J. The influence of clinical course after lung transplantation on rehabilitation success. Transpl Int. 2013 Mar;26(3):322-30. doi: 10.1111/tri.12048. Epub 2013 Jan 7. PMID 23294442